CLINICAL TRIAL: NCT06086119
Title: Quality of Life and Voice Perception in Patients Laryngoctomized Phonatory Wearers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: San Giovanni Addolorata Hospital (Other); Azienda Policlinico Umberto I (Other)
Responsible Party: Sponsor
Other Study IDs: RS1497/21
Record Dates: First submitted 2023-03-29; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-06

CONDITIONS: Quality of Life; Larynx Cancer
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who will be subjected to total laryngectomy and placement of voice prosthesis: Prospective, multicenter observational study involving patients who will be subjected to total laryngectomy and placement of voice prosthesis.Evaluate the patient's quality of life and voice perception underwent surgery for the placement of a voice prosthesis, through the administration of validated quality of life questionnaires: EORTC QLQ - H&N35; EORTC QLQ -C30, V-RQOL, VHI, SECEL3,4
  Interventions: Diagnostic Test: to assess the voice perception of the patient undergoing phonatory prosthesis placement surgery by evaluating the optimal score (>30) in terms of VHI.

INTERVENTIONS:
Diagnostic Test: to assess the voice perception of the patient undergoing phonatory prosthesis placement surgery by evaluating the optimal score (>30) in terms of VHI. — Prospective, multicenter observational study involving patients who will undergo total laryngectomy surgery and placement of phonatory prosthesis

SUMMARY:
Prospective, multicenter observational study involving patients who will undergo total laryngectomy surgery and placement of phonatory prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo laryngeal demolition surgery, total laryngectomy, who agree to phonatory prosthesis placement
* Patients who have undergone previous total laryngectomy surgery and intend to undergo placement of phonatory prosthesis.
* Age > 18 years
* Written informed consent

Exclusion Criteria:

* Patients who have not undergone demolitive surgical treatment by total laryngectomy or who do not accept the placement of phonatory prosthesis.
* Patients who are unable to complete questionnaires/follow the rehabilitation pathway

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Prospective, multicenter observational study involving patients who will undergo total laryngectomy surgery and placement of phonatory prosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2024-05-04 (Estimated)

PRIMARY OUTCOMES:
evaluate the patient's quality of life and voice perception underwent surgery for the placement of a voice prosthesis | Enlistment period: 2 years Total duration of the study: 36 months
  Evaluate the perception of the voice of the patient undergoing surgery of voice prosthesis positioning, evaluating the optimal score (>30) in terms of VHI.
  To calculate the sample size we based our estimate on the percentage of patients not undergoing voice prosthesis with a VHI score greater than 30 (Good Score). Such percentage is approximately 35%, a figure reported in the literature. Assuming a difference of 25% in terms of percentage of patients undergoing voice prosthesis who have a VHI score greater than 30 (60%) to ensure a power (1-β) equal to 80% and an α error of 5%, it will be necessary to enlist a total of 31 patients with the required requirements. Descriptive statistics will be calculated for all variables of interest. The associations will come evaluated using Fisher's exact test. Differences between subgroups will be assessed using the Mann-Whitney U test. All statistical analyzes were conducted using SPSS statistical software (version 21.0)

CONTACTS AND LOCATIONS:
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided